CLINICAL TRIAL: NCT02215577
Title: Comparison of Two Different Models of Liver Growth Stimulation in Advanced Colorectal Liver Metastatic Disease, (LIGRO Trial) Enabling Liver Resection
Brief Title: ALPPS Versus PVE/PL
Acronym: LIGRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regionalt Cancercentrum Väst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SweLiv 1-2014
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: cancer, colorectal; hepatectomy; portal vein; embolization; two-stage
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ligation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In-situ split with portal vein ligature (Experimental): In-situ liver split at time when portal vein ligature is performed
  Interventions: Procedure: In-situ split
- Portal embolization or ligation (Active Comparator): Intervention: Preoperative portal embolization (+/-ablation) followed by liver resection, or local resections and/or ablations followed by lobectomy, two-stage hepatectomy
  Interventions: Procedure: Portal embolization or ligation

INTERVENTIONS:
Procedure: In-situ split — The portal branches to the diseased side should be completely divided. The bile duct to the diseased side should not be divided. The parenchyma should be transected all the way through the transection plane and place a plastic sheet on the diseased transection surface.
  Other Names: ALPPS
  Arms: In-situ split with portal vein ligature
Procedure: Portal embolization or ligation — Portal vein embolization is performed according to the intervention used at the different sites.
  Arms: Portal embolization or ligation

SUMMARY:
Study Title Comparison of two different models of liver growth stimulation in advanced colorectal liver metastatic disease, (LIGRO Trial) enabling liver resection

Methodology Scandinavian Multiple Center Randomized Registry Based Clinical Trial

Study duration The planned duration of study participation for an individual subject from inclusion to follow-up are 3 years

Primary investigator:

Per Sandstrom (Linköping)

Number of subjects 100 patients randomized in a 1:1 randomization

Diagnosis and main inclusion criteria Patients with colorectal liver metastasis requiring liver resection, but are not resectable in one step because of a future liver remnant/standardized total liver volume of < 30 % extrahepatic metastatic disease is not an exclusion criteria if they can be addressed surgically in the future

Overall goal To evaluate if the ALPPS approach is superior to PVE in enabling patients, primarily unresectable due to inadequate FLR, to be resected and reach an R0 situation with an acceptable level of complications and perioperative mortality.

To evaluate if the ALPPS approach increases the growth rate of the liver compared to portal embolization or portal ligation leading to a shorter treatment period.

In addition the investigators aim to study if ALPPS may reach these goals without detectable or improved differences in tumor activity (PFS and OS), but with a shorter recovery and a higher proportion of patients reaching R0.

Hypothesis A higher proportion of patients can be resected with ALPPS counted as rate resected compared to the previously established methods with portal ligation or embolization.

This increased resection rate will not reduce the R0 rate, or increase the rate of Clavien grade 4 complication or higher (H0).

The ALPPS approach will increase the growth rate compared to portal embolization/ligation measured one week after the primary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. By liver tumor board found accepted for inclusion
2. Patients with a tumor burden of colorectal liver metastasis
3. Signed informed content
4. Colorectal liver metastatic disease with an estimated FLR/sTLV of <30%
5. Primary tumor and any extrahepatic disease possible to resect in patients with liver first approach or after resection of primary tumor.

Exclusion Criteria:

1. Cirrhosis
2. Significant comorbidity rendering subjects unsuitable for major surgery
3. Progressive disease after preoperative oncological treatment
4. Age<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate, the rate of liver resection in each study arm | 8 weeks
  For both the ALPPS and the portal vein embolization/ligation arm, resection is not allowed within the study if the patient is not reaching a future liver remnant of 30%.
  For both groups carcinomatosis or more metastases making aiming radical resections impossible will be seen as failures.

SECONDARY OUTCOMES:
Liver growth rate | At one week after primary intervention
  Liver growth is measured with regard to the future liver remnant by measuring the kinetic growth rate by performing repeated CT or MRI at one week after portal vein embolization/ligation or after the first step of the ALPPS procedure.

OTHER OUTCOMES:
Radical resection rate | 8 weeks
  Radical resection at resection line according to histopathology
Composite complication rate | 1 month after final surgery
  Overall complications will be analysed as a composite endpoint (CEP) including: ascites, postresectional liver failure, bile leak, intra abdominal bleeding, intraabdominal abscess and mortality, all with a Clavien score of at least 3
Treatment time | 8 weeks
  Treatment time in days from PVE/PL or date of ALPPS op 1 until date of leaving hospital after final surgery.
Progression free survival | 24 months
  Progression free survival according to randomization group.
Overall survival | Up to 24 months after last inclusion
  Overall survival after inclusion
Quality of life | 24 months post final resection
  Quality of life is measured by EORTC QLQ C-30 EQ5D ar 1,6,12,24 months.
Health economy | At 8 weeks
  An analysis with regard to hospitalisation rate and number of days in-ward between randomization arm.

CONTACTS AND LOCATIONS:
Locations (7):
- Departments of Surgical Gastroenterology and Transplantation, Copenhagen, Denmark
- Rikshospitalet Oslo University Hospital, Oslo, Norway
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Department of Surgery, Linkoping University Hospital, Linköping
  - Department of Surgery, University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Norrland University Hospital, Umeå

REFERENCES:
- [Derived] Hasselgren K, Rosok BI, Larsen PN, Sparrelid E, Lindell G, Schultz NA, Bjornbeth BA, Isaksson B, Larsson AL, Rizell M, Bjornsson B, Sandstrom P. Response to Comment on: Hasselgren K, et al ALPPS Improves Survival Compared With TSH in Patients Affected of CRLM: Survival Analysis From the Randomized Controlled Trial LIGRO. Ann Surg. 2021;273(3):442-448. Ann Surg. 2022 Nov 1;276(5):e632-e633. doi: 10.1097/SLA.0000000000005268. Epub 2021 Oct 20. No abstract available. PMID 35129514